CLINICAL TRIAL: NCT06099548
Title: First-in-Human (FIH) Clinical Investigation Protocol of the Magenta Elevate™ Percutaneous Left Ventricular Assist Device (pLVAD) System in Patients Undergoing Non-emergent, High-risk Percutaneous Coronary Interventions (ELEVATE I)
Brief Title: Magenta Elevate™ First-in-Human Clinical Study in High-Risk PCI Patients
Acronym: ELEVATE I
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Magenta Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRD00385
Record Dates: First submitted 2023-10-18; First posted 2023-10-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: High-Risk Percutaneous Coronary Intervention
Keywords: HR-PCI; High-risk percutaneous coronary intervention; Mechanical Circulatory Support; Left ventricular unloading; HRPCI; Temporary MCS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HR-PCI patients (Experimental): Patients undergoing non-emergent, high-risk percutaneous coronary interventions
  Interventions: Device: The Elevate™ System

INTERVENTIONS:
Device: The Elevate™ System — The Magenta Elevate™ is a temporary (≤ 6 hours) ventricular support device indicated for use during high-risk percutaneous coronary interventions (HR-PCI) performed electively or urgently in hemodynamically stable patients, with severe coronary artery disease.

SUMMARY:
The Elevate™ First-In-Human (FIH) study is designed to evaluate the initial safety and device functionality of the Elevate™ percutaneous Left Ventricular Assist Device (pLVAD) System in patients undergoing non-emergent, high-risk percutaneous coronary interventions.

DETAILED DESCRIPTION:
The Elevate™ System FIH study is planned as a prospective, single-arm, interventional study of up to 20 patients.

The Magenta Elevate™ is a temporary (≤ 6 hours) ventricular support device indicated for use during high-risk percutaneous coronary interventions (HR-PCI) performed electively or urgently in hemodynamically stable patients, with severe coronary artery disease.

The Magenta Elevate™ Pump is a catheter-mounted, self-expanding and retrievable pump, designed to unload the left ventricle by actively transporting blood from the left ventricle into the ascending aorta.

ELIGIBILITY:
Inclusion Criteria:

1. Non-emergent, percutaneous coronary intervention is planned in at least one stenotic lesion of a native coronary artery or bypass graft (de novo or restenosis)
2. Ejection fraction of ≤ 45% and at least one of the following:

   1. Intervention on an unprotected left main coronary artery
   2. Intervention on a last patent coronary conduit
   3. Three-vessel disease (in case of left coronary artery dominance, the combination of a Left Anterior Descending Artery (LAD) lesion and a proximal Left Circumflex Artery (LCX) lesion qualifies as three-vessel disease)
3. Femoral artery diameter compatible with the use of Elevate™
4. Subject signed informed consent

Exclusion Criteria:

1. Subject age < 40 or ≥ 83 years
2. Cardiogenic shock
3. Left ventricular mural thrombus
4. Presence of a mechanical aortic valve or a heart-constrictive device
5. Aortic stenosis
6. Moderate or severe aortic regurgitation (≥ 2+ by Transthoracic Echocardiography)
7. Severe peripheral vascular disease
8. Aortic pathology, such as aortic aneurysms, extreme tortuosity or calcifications that could pose an undue additional risk to the placement of a pLVAD device
9. Chronic renal dysfunction (serum creatinine ≥ 3.5 mg/dL)
10. Uncorrectable abnormal coagulation parameters (defined as platelet count ≤ 75,000 or INR ≥ 2.0 or fibrinogen ≤ 1.5 g/L)
11. Active systemic infection
12. Stroke or transient ischemic attack within 3 months of enrollment
13. Female subjects who are pregnant or breast-feeding

Ages: 40 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Device Performance | Through the end of the procedure
  Rate of procedural hypotension
Device Safety | Through the end of the procedure
  Rate of Major Device-Related Adverse Events

CONTACTS AND LOCATIONS:
Locations (2):
- Georgia (2):
  - Israeli-Georgian Medical Research Clinic "Helsicore", Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi